CLINICAL TRIAL: NCT04066322
Title: Resection of Metastatic Pancreatic Neuroendocrine Tumors After Induction System Treatment: Real World Study
Brief Title: Resection of Metastatic Pancreatic Neuroendocrine Tumors After Induction System Treatment
Acronym: RMPanNET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, Principal Investigator, Fudan University
Other Study IDs: CSPAC-26
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Neuroendocrine Tumors; Metastases; Surgery
MeSH Terms: conditions — Neuroendocrine Tumors; Neoplasm Metastasis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- system treatment: Patients continue to receive standard system treatment, including SSA, targeted therapy and chemotherapy.
  Interventions: Other: system treatment
- system treatment and Surgery: Patients receive synchronous resection of primary tumor and metastasis after system treatment. and treatment after surgery is based on the clinical decision.
  Interventions: Procedure: system treatment and surgery

INTERVENTIONS:
Procedure: system treatment and surgery — to patients with PR/SD after system treatment, investigator assess the tumor is resectable, and participants decide to receive Synchronous resection of primary tumor and metastasis. after surgery, the investigator decide further treatments.
  Other Names: resection of primary and metastatic tumors
  Groups: system treatment and Surgery
Other: system treatment — to patients with PR/SD after system treatment, investigator assess the tumor is resectable, and participants decide to continue take system treatment.
  Groups: system treatment

SUMMARY:
This study is to evaluate the efficacy and tolerability of surgery in selecting patients who can benefit from the synchronous resection of primary pancreatic neuroendocrine tumor and liver metastasis after induction systemic treatment. The willing of participants decide who receive surgery and who will continue to receive standard systemic treatment.

DETAILED DESCRIPTION:
system treatments of metastatic PanNET include SSA, sunitinib, mTOR inhibitor and chemotherapy. For patients achieved PR/SD after system treatment, resection of primary tumor and metastasis maybe a better way to decline tumor burden and get longer survival. this real world study is focused on this group of patients with metastatic PanNET, and to evaluate the efficacy and tolerability of surgery in selecting patients who can benefit from the synchronous resection of primary pancreatic neuroendocrine tumor and liver metastasis after induction systemic treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy-proven neuroendocrine tumor
2. primary site in pancreas
3. Advanced disease with lymph node or distant metastases (N1, M1) cannot undergoing cytoreduction by surgery/local ablative therapy at the diagnosis
4. curative intent of all therapies possible
5. ECOG 0-2

Exclusion Criteria:

1. Undifferentiated neuroendocrine carcinoma or mixed neuroendocrine carcinoma secondary tumor
2. functioning NET or advanced carcinoid heart disease
3. part of hereditary syndrome, such as MEN1, VHL
4. do not willing to receive systemic treatment
5. diagnosed with other cancer within 5 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with metastatic pancreatic neuroendocrine tumors in a tertiary referal center
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-08-25 (Actual); Primary Completion 2024-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 5 years

SECONDARY OUTCOMES:
overall survival | 5 years
Number of Postoperative morbidity | Up to 90 days after operation
  Including pancreatic fistula, biliary fistula, hemorrhage, wound infection, delayed gastric emptying, reoperation
number of Postoperative mortality | Up to 90 days after operation

OTHER OUTCOMES:
number of Patients die from any cause during 90 days after operation | 5 years
progression-free survival in subgroup analysis | 5 years
  liver metastasis type, grade, extrahepatic metastasis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No